CLINICAL TRIAL: NCT00678366
Title: Evaluation of Adding Small Amounts of Oxygen to the CO2 Pneumoperitoneum Upon Pain and Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Jasper Verguts, MD, PhD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PK-001
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Pain; Inflammation
Keywords: laparoscopy; carbon dioxide; oxygen; pain; inflammation
MeSH Terms: conditions — Pain; Inflammation | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): addition of 4% oxygen to the carbon dioxide pneumoperitoneum
  Interventions: Procedure: addition of 4% oxygen
- 2 (Active Comparator): pure carbon dioxide pneumoperitoneum
  Interventions: Procedure: carbon dioxde

INTERVENTIONS:
Procedure: addition of 4% oxygen — addition of 4% oxygen to the carbon dioxide pneumoperitoneum
  Arms: 1
Procedure: carbon dioxde — classic pneumoperitoneum with 100 % carbon dioxide
  Arms: 2

SUMMARY:
The study intends to investigate the use of a novel gaz-composition used during laparoscopy upon pain and inflammation in the post-operative period.

DETAILED DESCRIPTION:
Laparoscopic surgery was introduced by gynaecologists in a search for a minimally invasive surgical approach. Laparoscopy is now generally accepted and widely used in different medical fields (gynaecology, digestive surgery, oncology, etc.,.).

1. CO2 pneumoperitoneum and pain:

   Carbon dioxide is generally used to induce and maintain a pneumoperitoneum. Following a diagnostic procedure post-operative pain is generally low. For more extensive laparoscopic surgery, pain is related to the type of surgery. It has been suggested that pain also increases with the duration of surgery.
2. CO2 pneumoperitoneum and inflammation Different immune mediators were already evaluated during laparoscopic surgery. On peripheral blood interleukin-6, C-reactive protein, tumor necrosis factor, interleukin-1, histamine response, total leukocyte counts and T-lymphocyte populations, delayed-type hypersensitivity and neutrophils activation and function were evaluated. Local peritoneal host defences such as macrophage activation and function and leukocyte function have also been studied.

   Laparoscopic surgery is associated with less post-operative inflammatory reaction and less immune activation then laparotomy. (1-2).

   The degree of alteration in C-reactive proteins was noted to be a 5 fold increase after laparoscopic cholecystectomy (3).

   Peripheral leukocyte populations may not be the principal determinant of an acute-phase response as much as an hepatic response to stress and injury. Kloosterman (4) has demonstrated a transient increase in granulocyte numbers after open cholecystectomy but not after laparoscopic cholecystectomy.

   Interleukin-6 levels have been noted to be reduced in patients undergoing laparoscopic procedures compared to traditional laparotomy, with a linear correlation between peak concentrations of IL-6 and C-reactive proteins (3).

   West (5) investigated the production of cytokines in peritoneal macrophages incubated in carbon dioxide. Macrophage TNF and IL-1 responses to bacterial endotoxin were lower for macrophages incubated in carbon dioxide than in either air or helium. A proposed mechanism for this difference was that carbon dioxide affected the intracellular medium by creating a more acidic environment. He speculates that the impairment in peritoneal macrophage cytokine production may contribute to an apparent lack of inflammatory systemic response during laparoscopic surgery rather than the physiologic stress of the surgery itself. This provides a potential molecular mechanism to explain peritoneal macrophage immunosuppression.
3. Effects of adding 2-4 % of oxygen to the CO2 pneumoperitoneum Adding 4% of oxygen to the CO2 results in a partial oxygen pressure of 30 mmHg (4% of 760 atmospheric pressure + 15 mmHg insufflation pressure) which is similar to the physiologic 20-40 mmHg partial oxygen pressure for peripheral tissues.

   In a series of experiments it was demonstrated that adhesion formation decreased by 50% when 0.7-1% of oxygen was added to the CO2 pneumoperitoneum. Adding 2-4% of oxygen to the CO2 pneumoperitoneum completely prevented this effect. This observation is consistent with the oxygen tensions known to induce hypoxia inducible factor (HIF) and with the normal physiologic peripheral partial oxygen tension around 20-40 mm Hg. (6) In addition, CO2 resorbtion was profoundly affected by adding 2-4% of oxygen in our rabbit model. (7) From these studies we concluded that during CO2 pneumoperitoneum the progressively increasing resorbtion of CO2 is completely prevented by adding 2-4% of oxygen.
4. Pneumoperitoneum and the mesothelial barrier The effect of pneumoperitoneum upon CO2 resorbtion and adhesion formation are consistent with mesothelial hypoxia. This hypoxia causes the large, flat mesothelial cells to retract and bulge thus exposing increasingly large areas of extra cellular matrix (ECM) in between the cells as demonstrated in mice and rats. (8) This moreover may facilitate malignant tumor implantation. Where it has been suggested to affect adversely intraperitoneal infections. (9-11)
5. Insufflation with oxygen We will use a premixed bottle of CO2 + 4% oxygen to insufflate the abdomen. The mixture is stable.

4 % of oxygen obviously does not cause an electrosurgical risk since air contains 20% of oxygen. Also the eventual accidental intravenous perfusion of 1L min would result in the perfusion of 0.04 L/min of oxygen which is considered harmless.

Hypothesis:

We assume that decreasing the hypoxic damage to the mesothelium by adding 4% of oxygen to the CO2 pneumoperitoneum will decrease the inflammatory reaction and therefore post-operative pain and faster normalisation of inflammation parameters.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed a written informed consent to participate in the study and has agreed to follow instructions and complete all required questionnaires
* Females, 18 years of age or older
* She has to undergo a planned laparoscopy for mentioned indications with a duration that exceeds 60 minutes

Exclusion Criteria:

* Pregnancy
* Immunodeficiency
* Refuse or unable to sign informed consent
* Chronic diseases (i.e. COPD, Crohn, cardiac…)
* Mental diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
to check if the post-operative pain and inflammatory reaction after laparoscopy decreases when CO2 with the addition of 4% of oxygen is used instead of pure CO2 | 1 week

SECONDARY OUTCOMES:
the effects on CO2 resorbtion, pain and inflammation by co-variables: body mass index, length of surgery, painkiller intake and pain before surgery as defined by the Biberoglu and Behrman scale | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Koninckx, MD, PhD, Principal Investigator — UZ Leuven, campus Gasthuisberg
Locations (1):
- UZ Leuven, campus gasthuisberg, Leuven, Vlaams Brabant, Belgium